CLINICAL TRIAL: NCT00667563
Title: A Single-Arm, Open-Label Pilot Study of the Safety and Immunogenicity of the Merck Quadrivalent Human Papillomavirus Vaccine Among HIV-Positive Women in India
Brief Title: Vaccine Therapy in Preventing HPV in HIV-Positive Women in India
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AMC-054; U01CA121947 (NIH); CDR0000593634 (Other: NCI)
Record Dates: First submitted 2008-04-25; First posted 2008-04-28 (Estimated); Results first posted 2014-04-11 (Estimated); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Cervical Cancer; Nonneoplastic Condition; Precancerous Condition
Keywords: human papilloma virus infection; cervical cancer; cervical intraepithelial neoplasia; HIV infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Papillomavirus Infections; Uterine Cervical Dysplasia; HIV Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Gardasil Vaccination (Experimental): Vaccination with the Quadrivalent Human Papillomavirus Recombinant vaccine (0.5 mL Gardasil®) by intramuscular (IM) injection at Day 0, Weeks 8 and 24.
  Interventions: Biological: quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine; Genetic: DNA analysis; Genetic: polymerase chain reaction; Other: cytology specimen collection procedure; Procedure: colposcopic biopsy

INTERVENTIONS:
Biological: quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine — Vaccination with the Quadrivalent Human Papillomavirus Recombinant vaccine (0.5 mL Gardasil®) by intramuscular (IM) injection at Day 0, Weeks 8 and 24.
Genetic: DNA analysis — Weeks 0, 2, 10, 26, and 52.
  Other Names: HIV viral load test and HPV neutralization assays.
Genetic: polymerase chain reaction — Screening, week 36, and week 52.
Other: cytology specimen collection procedure — Screening, week 36, and week 52.
Procedure: colposcopic biopsy — Screening, week 36, and week 52.

SUMMARY:
RATIONALE: Vaccines made from virus proteins may help the body build an effective immune response to prevent cervical cancer.

PURPOSE: This pilot study is looking at the side effects of a human papillomavirus vaccine and how well it works in preventing cervical cancer in women in India with HIV-1 infection.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the safety of the Gardasil® quadrivalent human papillomavirus (HPV) (types 6, 11, 16,18) virus-like-particle vaccine with vs without prior exposure to one or more of the HPV types in the vaccine in HIV-positive women in Chennai, India.
* Determine the effect of the vaccine on HIV viral load and CD4+/CD8+ levels in these patients.
* Determine the proportion of these patients who respond serologically to the HPV vaccine and the kinetics of their response.

Secondary

* Determine the prevalence and incidence of cervical intraepithelial neoplasia in these patients.
* Determine the spectrum of cervical HPV types in these patients at baseline, 9 months, and 1 year after vaccination.

OUTLINE: This is a multicenter study.

Patients receive quadrivalent human papillomavirus (HPV) (types 6, 11, 16, 18) recombinant vaccine intramuscularly on day 0 and once in weeks 8 and 24.

Patients undergo cervical cell, buccal cell, and blood sample collection at baseline and periodically after vaccination for immunologic and virologic studies. Cervical cytology specimens are examined by polymerase chain reaction to detect HPV 6, 11, 16, or 18 DNA, as well as 35 other HPV types. Blood samples are analyzed for CD4+/CD8+ cell count, plasma HIV-1 RNA levels, and serum HPV antibody titers for HPV types 6, 11, 16, and 18. Some plasma samples will be stored for future HPV pseudovirion neutralization assays.

After completion of study therapy, patients are followed periodically for up to 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* HIV-1 infection, as documented by any licensed ELISA test kit and confirmed by western blot before study entry

  * HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test
* Meets 1 of the following criteria:

  * Nadir CD4 level of ≤ 350 cells/mm³ and receiving highly active antiretroviral therapy (HAART) for at least 6 months before study entry
  * Nadir CD4 level of > 350 cells/mm³ and not receiving HAART at the time of study entry
* No known history of high-grade CIN or cervical cancer

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* ANC > 750 cells/mm³
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100,000/mm³
* Serum creatinine ≤ 3 times upper limit of normal (ULN)
* AST and ALT ≤ 3.0 times ULN
* Conjugated (direct) bilirubin ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active drug or alcohol use or dependence that would interfere with adherence to study requirements, in the opinion of the site Investigator
* No serious illness requiring systemic treatment and/or hospitalization within the past 45 days
* No allergy to yeast or any of the components of quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 45 days since prior systemic antineoplastic or immunomodulatory treatment, systemic corticosteroids, investigational vaccines, interleukins, interferons, growth factors, or intravenous immunoglobulin

  * Routine standard of care, including hepatitis B, influenza, and tetanus vaccines are allowed

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Palefsky, MD, Study Chair — University of California, San Francisco; N. Kumarasamy, MD, Principal Investigator — YRG Care
Locations (1):
- YRG Care, Chennai, India

REFERENCES:
- See also: Clinical trial summary for AMC-054 — https://clinicaltrials.gov/study/NCT00667563

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gardasil Vaccination
Started | 150
Completed | 126
Not Completed | 24
Not completed — Protocol Violation | 24

BASELINE CHARACTERISTICS:
Population: Enrolled in study
Arm/Group | Gardasil Vaccination
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety, in Terms of Grade 3 or 4 Adverse Events Attributed to the Vaccine, According to NCI CTCAE v3.0
Description: Number of grade 3 or 4 adverse events attributed to vaccine per 100 patients
Time Frame: 52 weeks from study entry
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: Grade 3/4 adverse events per 100 patient
Arm/Group | Gardasil Vaccination
Number analyzed (Participants) | 150
Grade 3/4 adverse events per 100 patient | 6.0 [3.12 to 11.58]

2. Primary Outcome: Number of Patients With Significant Decrease (at the 0.05 Significance Level) in CD4+ Cell Count
Description: Significant decrease (at the 0.05 significance level) in CD4+ cell count to 75% of the baseline level on two or more consecutive tests
Time Frame: Screening/Week 0, Weeks 2, 10, 26, and 52.
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Gardasil Vaccination
Number analyzed (Participants) | 150
participants | 11 [3.77 to 12.91]

3. Primary Outcome: Number of Patients With Detectable HPV Antibodies to HPV 16 at Week 28
Description: Number of participants with detectable HPV antibody to HPV 16 among those with undetectable antibodies to HPV 16 at baseline
Time Frame: Week 28
Population: Per-protocol population with undetectable HPV-16 levels at baseline
Measure: Number; unit: participants
Arm/Group | Gardasil Vaccination
Number analyzed (Participants) | 96
participants | 95

4. Primary Outcome: Number of Patients With a Significant Increase in HIV Viral Load
Description: Number of patients with a significant increase in HIV viral load defined as > 1 log increase in HIV load from baseline on 2 consecutive occasions
Time Frame: Screening/week 0, weeks, 2, 10, 26 and 52
Measure: Number; unit: participants
Arm/Group | Gardasil Vaccination
Number analyzed (Participants) | 150
participants | 7 [1.95 to 9.63]

5. Primary Outcome: Number of Patients With Detectable Antibodies to HPV-6
Description: Detectable antibodies to HPV-6 among participant who had undetectable antibodies to HPV-6 at baseline
Time Frame: 28 weeks
Population: Per-protocol participants with undetectable antibodies to HPV-6 at baseline
Measure: Number; unit: participants
Arm/Group | Gardasil Vaccination
Number analyzed (Participants) | 88
participants | 88

6. Primary Outcome: Number of Patients With Detectable Antibodies to HPV-11
Description: Detectable antibodies to HPV-11 among those who had undetectable antibodies to HPV-11 at baseline
Time Frame: 28 weeks
Population: Per-protocol population of participants with undetectable antibodies for HPV-11 at baseline
Measure: Number; unit: participants
Arm/Group | Gardasil Vaccination
Number analyzed (Participants) | 111
participants | 110

7. Primary Outcome: Number of Patients With Detectable Antibodies to HPV-18
Description: Detectable antibodies to HPV-18 among participants with undetectable antibodies to HPV-18 at baseline
Time Frame: 28 weeks
Population: Per-protocol population of participants with undetectable HPV-18 antibodies at baseline
Measure: Number; unit: participants
Arm/Group | Gardasil Vaccination
Number analyzed (Participants) | 104
participants | 94

ADVERSE EVENTS:
Arm/Group | Gardasil Vaccination
Serious Adverse Events (participants affected / at risk) | 4/150
Other Adverse Events (participants affected / at risk) | 145/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gardasil Vaccination (N=150)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Leptospirosis (Infections and infestations) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gardasil Vaccination (N=150)
Abdominal pain (Gastrointestinal disorders) | 35 (41)
Dyspepsia (Gastrointestinal disorders) | 19 (22)
Vomiting (Gastrointestinal disorders) | 10 (11)
Fatigue (General disorders) | 27 (32)
Lung Infection (Infections and infestations) | 8 (8)
Skin Infection (Infections and infestations) | 26 (29)
Upper Respiratory Infection (Infections and infestations) | 44 (60)
Vaginal Infection (Infections and infestations) | 21 (22)
Vulval Infection (Infections and infestations) | 10 (10)
Anorexia (Metabolism and nutrition disorders) | 21 (24)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (40)
Myalgia (Musculoskeletal and connective tissue disorders) | 25 (34)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 45 (61)
Headache (Nervous system disorders) | 34 (47)
Vaginal Discharge (Reproductive system and breast disorders) | 21 (27)
Cough (Reproductive system and breast disorders) | 59 (87)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 (22)
Pruritus (Skin and subcutaneous tissue disorders) | 41 (64)
Rash, maculo-papular (Skin and subcutaneous tissue disorders) | 14 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No